CLINICAL TRIAL: NCT00846963
Title: Ursodiol for Treating Parenteral Nutrition Associated Cholestasis in Neonates
Acronym: URSONEONAT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ibrahim Mohamed (Other)
Responsible Party: Sponsor-Investigator, Ibrahim Mohamed, Assisstant professor of pediatrics, St. Justine's Hospital
Organization: St. Justine's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RC:127
Record Dates: First submitted 2009-02-17; First posted 2009-02-19 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Cholestasis
Keywords: parenteral nutrition associated cholestasis in neonates; parenteral nutrition induced cholestasis in preterms; Bile duct obstruction; biliary stasis
MeSH Terms: conditions — Cholestasis | interventions — Ursodeoxycholic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ursodiol (Experimental): Participants assigned in this arm receive an ursodiol suspension at 20mg/ml.
  Interventions: Drug: Ursodiol
- placebo (Placebo Comparator): A placebo suspension that looks like the ursodiol suspension used.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Ursodiol — Ursodiol is given by mouth, three times a day from second value of elevated conjugated bilirubin (>33mmol/L) to the resolution of cholestasis (conjugated bilirubin <34mmol/L) If Nil per os, 3,3mg/kg/dose is given. If Nil per os is required (e.g. pre-surgery, or necrotizing enterocolitis), none is given.
  If enteral feeding is under 100mL/kg/day, 6,7 mg/kg/day is given. If enteral feeding exceeds 100mL/kg/day, 10 mg/kg/day is given.
  Other Names: Urso; ursodeoxycholic acid
  Arms: Ursodiol
Drug: placebo — Placebo given in the same amount that ursodiol would be given, depending on enteral feeding and weight. It is also given three times a day, until cholestasis resolution.
  Arms: placebo

SUMMARY:
The purpose of this study is to determine whether ursodiol is effective in the treatment of parenteral nutrition associated cholestasis in neonates.

DETAILED DESCRIPTION:
This is the first randomised controlled study that address the question of the role of ursodiol as treatment of cases of PNAC.

It includes all neonates with stratification of less than and equal to 32 weeks or more than 32 weeks of gestation.

ELIGIBILITY:
Inclusion Criteria:

* Preterm or in-term newborns hospitalized in neonatal care units at CHU Sainte-Justine between October 1st 2008 and October 1st 2011.
* Must be receiving parenteral nutrition (either partial or total) at the diagnosis of cholestasis.
* Parental Consent must be obtained.

Exclusion Criteria:

* Active urinary tract infection
* Presence of clinical signs(acholic stool) of or ultrasound evidence of biliary tract anomalies.
* Positive TORCH infections(Toxoplasmosis, Other infections, Rubella, Cytomegalovirus, Herpes simplex virus)
* Known short bowel syndrome
* Known congenital hypothyroidism
* Known genetic disorders associated with cholestasis like galactosemia, phenylcytonuria, antitrypsin 1 deficiency... etc

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2008-10; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Length of parenteral nutrition associated cholestasis (in days) | at the end of cholestasis (when conjugated bilirubin < 34 mmol/L) average of 4 weeks.

SECONDARY OUTCOMES:
Peak value of biomarkers associated with cholestasis (Gamma-glutamyl transpeptidase, Alkaline phosphatase, conjugated bilirubin) | at least once a week, during cholestasis
1- Other hepatic marker (Aspartate transaminase, alanine transaminase, albumin blood level) | at least once a week, during cholestasis
Length required to minimal enteral feeding (120mL/kg/day) measured in days. | From birth to outcome (usually less than 21 days)
Weight gain (in g/kg/day) | From birth to resolution of cholestasis (very varuiable but usually less than 3 months)
Adverse effects linked to ursodiol | From beginning to the end of the medication (average 4 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim Mohamed, MB ChB, DIS P, Principal Investigator — St. Justine's Hospital; Josianne Malo, B.Pharm, M.Sc., Study Director — St. Justine's Hospital
Locations (1):
- CHU Sainte-Justine, Montreal, Quebec, Canada

REFERENCES:
- [Background] Al-Hathlol K, Al-Madani A, Al-Saif S, Abulaimoun B, Al-Tawil K, El-Demerdash A. Ursodeoxycholic acid therapy for intractable total parenteral nutrition-associated cholestasis in surgical very low birth weight infants. Singapore Med J. 2006 Feb;47(2):147-51. PMID 16435058
- [Background] Arslanoglu S, Moro GE, Tauschel HD, Boehm G. Ursodeoxycholic acid treatment in preterm infants: a pilot study for the prevention of cholestasis associated with total parenteral nutrition. J Pediatr Gastroenterol Nutr. 2008 Feb;46(2):228-31. doi: 10.1097/MPG.0b013e3181560524. PMID 18223390
- [Background] Chen CY, Tsao PN, Chen HL, Chou HC, Hsieh WS, Chang MH. Ursodeoxycholic acid (UDCA) therapy in very-low-birth-weight infants with parenteral nutrition-associated cholestasis. J Pediatr. 2004 Sep;145(3):317-21. doi: 10.1016/j.jpeds.2004.05.038. PMID 15343182
- [Background] Venigalla S, Gourley GR. Neonatal cholestasis. Semin Perinatol. 2004 Oct;28(5):348-55. doi: 10.1053/j.semperi.2004.09.008. PMID 15686266
- [Background] McKiernan PJ. Neonatal cholestasis. Semin Neonatol. 2002 Apr;7(2):153-65. doi: 10.1053/siny.2002.0103. PMID 12208100